CLINICAL TRIAL: NCT06537804
Title: Project Lung Cancer Screening in Southern Denmark
Acronym: PLUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: S-20240033
Record Dates: First submitted 2024-07-01; First posted 2024-08-05 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Low-dose CT scans are performed once a year from 2024 to 2026 to screen for lung cancer including a lung function test the first year of attendance (2024).
  Interventions: Radiation: Screening by low-dose CT scan
- Control (No Intervention): Citizens from the cohort who are randomized to no intervention.

INTERVENTIONS:
Radiation: Screening by low-dose CT scan — Screening for lung cancer by low-dose CT scan
  Arms: Intervention

SUMMARY:
One thousand randomly selected voluntary citizens aged 60-74 years old, who are heavy current or former smokers with an increased risk of developing lung cancer may be included in the project. The participants will be identified through an initial questionnaire survey concerning smoking history and general health. Project participants are offered a low-dose CT (LDCT) scan annually for three consecutive years. In relation to the first scan, a lung function test will also be performed. The screening process will be evaluated for possible national implementation of a lung cancer screening program in Denmark.

DETAILED DESCRIPTION:
This pilot study is a prospective interventional feasibility study. The primary goal is to evaluate the impact on healthcare organization, administration of resources and costs, and thereby assessing the feasibility of implementing systematic screening for lung cancer among people at high risk in Denmark (current or former heavy smokers). The pilot study will be performed on Funen in the Region of Southern Denmark and will run over three years (2024-2026). One thousand randomly selected participants aged 60-74 years old, who meet the screening criteria, will receive annual LDCT scans for three consecutive years.

Data will be collected continuously throughout the study period. The analysis method will focus on descriptive statistics to display questionnaire response and participation rates, and assess the impact of screening on healthcare organization and resources. Furthermore, the result including direct and indirect effects of the screening process (e.g. number of positive findings, false positive results, and follow-up rates). The analyses will also include healthcare economics including resource consumption as well as qualitative assessments to describe potential differences between the screening population versus a corresponding control group of heavy smokers. Finally, the radiologists' assessments of the project's LDCT scans are compared to the assessment of an artificially intelligent algorithm to explore the opportunities of supporting a future national screening program.

ELIGIBILITY:
Inclusion Criteria:

* Heavy smokers (≥ 30 pack years) or citizens with a PLCOm2012 calculated 6-year risk of lung cancer > 2%.
* Age: 60-74 years old
* Residence on Funen and surrounding islands

Exclusion Criteria:

* Cancer treatment or follow-up (except non melanoma skin cancer and similar low malignant cancers) within the past 12 months
* CT scan performed within the past 12 months

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1332 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung cancer screening cost-effectiveness analysis quantified in the form of incremental cost-effectiveness ratio threshold | Up to 36 months
  ratio

SECONDARY OUTCOMES:
Characteristics of citizens from the cohort based on registry data | Up to 36 months
  Registry data
Participation rate | 36 months (complete study period)
  Number and percentage of citizens completing the screening trial
Dropouts | 36 months (complete study period)
  Number and percentage of citizens included that dropout during the study period
Lung cancer found on low dose CT-scans | Baseline, after 1 year, after 2 years
  Number and percentage
Inconclusive or non-malignant findings on low dose CT scans | Baseline, after 1 year, after 2 years
  Number and percentage
FEV1 | Baseline
  Measured in liters by a lung function test
FVC | Baseline
  Measured in liters by a lung function test
Treatment diagnose - cancer | 36 months (complete study period)
  number and percentage of treatments by action diagnosis related to cancer
Hospitalization time | 36 months (complete study period)
  Hospitalization time related to lung cancer diagnosis measures in days
Treatment diagnose - any other disease (found on low dose CT scans) | 36 months (complete study period)
  number and percentage of treatment diagnosis related to findings of other diseases (by action diagnosis)
Referral to follow-up procedures | 36 months Entire study period
  Number of referrals
Self reported health and quality of life assessed by the EQ-5D-5L questionnair | Baseline and after 2 years
  level of percieved problems are coded from level 1 to 5 in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression"
Self-reported smoking status | Baseline, after 1 year, after 2 years
  Yes/no/former smoker
All-cause-mortality | 36 months (the entire study period)
  Number of deaths in both groups (intervention/no intervention)
Gender | Baseline
  Male/female
Weight | Baseline
  Kilogram
Height | Baseline
  Centimeters
Smoking history | baseline
  according to the PLCOm2012 risk model
Total time consumption of extra work at involved departments: department of lung diseases, department of radiology and department og pulmonary diseases | 36 months
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stenger, Consultant, Study Director — Odense University Hospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense, Region Syddanmark
  - Department of Radiology, Svendborg Hospital, Svendborg, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No